CLINICAL TRIAL: NCT03972969
Title: Highly Challenging Balance Program to Reduce Fall Rate in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E3055-R
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Exercise therapy; Accidental falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-person exercise group (Experimental): facility-based structured exercise program
  Interventions: Behavioral: Facility-based structured exercise
- Remote exercise group (Experimental): home-based structured exercise program
  Interventions: Behavioral: Home-based structured exercise
- Control group (Active Comparator): health education
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Facility-based structured exercise — Structured exercise program in a facility with instruction and encouragement
  Arms: In-person exercise group
Behavioral: Home-based structured exercise — Structured exercise program in the home with instruction and encouragement
  Arms: Remote exercise group
Behavioral: Health education — Provision of general information about a variety of topics
  Arms: Control group

SUMMARY:
This study will test the hypothesis that two highly challenging exercise programs, one based at the VA medical center and the other conducted remotely, will both significantly reduce overall fall rates in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background/Rationale. Parkinson's disease (PD) is the second most common neurodegenerative disease, affecting over one million Americans. The cardinal clinical manifestations of PD include resting tremor, rigidity, bradykinesia, and postural instability/gait disturbance. In addition, people with PD fall frequently, with 60% falling annually and two-thirds of these falling recurrently. Identifying interventions that successfully improve postural control and reduce fall rate is critical to reduce disability, improve quality of life, and potentially increase survival in patients with PD. Recent randomized, controlled trials (RCT) have examined the effects of exercise and physical therapy interventions on reducing falls in patients with PD; however, with mixed results.

Objectives. There is a limited availability of effective treatment options to reduce falls in PD. In this context, some studies suggest that highly challenging exercise approaches may lead to better outcomes. The investigators propose investigating the effects of two theoretically driven, progressive, highly challenging exercise programs: 1) a structured exercise program at the VA and 2) a structured exercise program at home. There will also be a control group in which health education is provided.

Methods. The investigators propose to conduct an RCT evaluating effects on fall rate. A total of 162 VA patients with mild-to-moderate PD will be randomly assigned to one of the three 3-month interventions: in-person exercise at the VA, remotely-delivered exercise, or health education. Outcomes will be compared between each intervention group and the control group. Fall rates will be compared between groups with the use of negative binomial regression models.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of idiopathic PD
* At least 2 of the 3 cardinal signs of PD (resting tremor, rigidity, bradykinesia)
* Response to dopaminergic medication

Exclusion Criteria:

* Angina pectoris
* History of myocardial infarction (MI) within 6 months
* History of ventricular dysrhythmia requiring current therapy

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886

RESULTS

PARTICIPANT FLOW:
Period: 3-month Follow-up
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group
Started | 51 | 58 | 53
Completed | 50 | 57 | 53
Not Completed | 1 | 1 | 0
Not completed — Death | 1 | 1 | 0
Period: 6-month Follow-up
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group
Started | 50 | 57 | 53
Completed | 47 | 54 | 50
Not Completed | 3 | 3 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group | Total
Number analyzed (Participants) | 51 | 58 | 53 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (7.0) | 76.2 (7.2) | 73.2 (7.7) | 74.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 51 | 57 | 52 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 51 | 58 | 51 | 160
  Race/Ethnicity: Black or African American | 0 | 0 | 1 | 1
  Race/Ethnicity: Hispanic or Latino | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Falls Over 3 Month Period
Description: Total number of falls from baseline to the 3-month follow-up. Falls are defined as unexpected events in which the participants come to rest on the ground, floor, or lower level.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: number of falls
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group
Number analyzed (Participants) | 51 | 58 | 53
number of falls | 1.1 (2.7) | 1.6 (3.0) | 9.7 (48.4)
Statistical Analysis 1: Comparison: In-person Exercise Group vs Control Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.13, 95% CI 2-sided [0.05 to 0.32]
Statistical Analysis 2: Comparison: Remote Exercise Group vs Control Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.25, 95% CI 2-sided [0.10 to 0.61]
Statistical Analysis 3: Comparison: In-person Exercise Group vs Remote Exercise Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.52, 95% CI 2-sided [0.19 to 1.38]

2. Secondary Outcome: Number of Falls Over 6 Month Period
Description: Total number of falls from baseline to the 6-month follow-up. Falls are defined as unexpected events in which the participants come to rest on the ground, floor, or lower level.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: number of falls
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group
Number analyzed (Participants) | 51 | 58 | 53
number of falls | 2.08 (3.46) | 3.02 (6.32) | 11.36 (49.55)
Statistical Analysis 1: Comparison: In-person Exercise Group vs Control Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.15, 95% CI 2-sided [0.07 to 0.33]
Statistical Analysis 2: Comparison: Remote Exercise Group vs Control Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.26, 95% CI 2-sided [0.11 to 0.58]
Statistical Analysis 3: Comparison: In-person Exercise Group vs Remote Exercise Group; Test type: Superiority; p < 0.05, negative binomial regression; Incidence Rate Ratio = 0.58, 95% CI 2-sided [0.25 to 1.38]

ADVERSE EVENTS:
Time Frame: Adverse events collected over the 6-month participation period
Arm/Group | In-person Exercise Group | Remote Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/51 | 2/58 | 1/53
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/58 | 0/53
Other Adverse Events (participants affected / at risk) | 0/51 | 0/58 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03972969/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03972969/ICF_000.pdf